CLINICAL TRIAL: NCT03787381
Title: Factors Influencing the Development of Uterine Niche After Cesarean Delivery
Brief Title: Uterine Niche After Cesarean Section
Acronym: AMSRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5562-18-SMC
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Uterine Scar From Previous Cesarean Delivery (Diagnosis)
Keywords: cesarean section, niche, uterine scar defect
MeSH Terms: conditions — Disease | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Uterine scar will be evaluated by vaginal ultrasound examination
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Vaginal ultrasound examination

SUMMARY:
In the past decade several articles have described a defect that can be seen on ultrasound at the site of cesarean delivery scar, known as a 'niche' .An incompletely healed scar is a long-term complication of cesarean delivery and is associated with symptoms such as postmenstual spotting, dysmenorrhoea, chronic pelvic pain dyspareunia and subfertility. This study aimes to evaluate the prevalence of niche in a large cohort study after long term follow up since operation, and characterize the risk factors for its development and for symptoms to appear.

DETAILED DESCRIPTION:
As the rate of cesarean deliveries continues to increase, concern regarding the association between delivery by cesarean section and long-term maternal morbidity has been growing . In the past decade several articles have described a defect that can be seen on ultrasound at the site of the cesarean delivery scar, known as a 'niche' .A 'niche' describes the presence of a hypoechoic area within the myometrium of the lower uterine segment, reflecting a discontinuation of the myometrium at the site of a previous cesarean delivery . An incompletely healed scar is a long-term complication of cesarean delivery and is associated with symptoms such as postmenstual spotting, dysmenorrhoea, chronic pelvic pain dyspareunia and subfertility.

The reported prevalence of a niche in non-pregnant women varies depending on the criteria used to define a niche, the time of evaluation since operation, method of detection, and study population. Osser et al. used the definition 'any visible defect' , Bij de Vaate et al. used 'any indentation of at least 1 mm and van der Voet used a cut-off level of 2 mm, however, consensus on the exact cut-off levels is lacking. As approximate evaluation to the operation, the prevalence reported is higher, as early scanning may facilitate the recognition of the location of the caesarean delivery scar in the uterine wall due to incomplete scar healing, with no definition of the most appropriate time since operation. Commonly used methods to evaluate the presence of a niche are trans vaginal ultrasound, sonohysterography and hysteroscopy with detection rate of approximately ~50% of women with previous cesarean section in all methods with no definition of the gold standard.

The aim of this study in to evaluate the prevalence of niche in a large cohort study after long term follow up since operation and characterize the risk factors for its development and for symptoms to appear.

ELIGIBILITY:
Inclusion Criteria:

* Women after cesarean delivery
* Minimum interval of 3 months since operation

Exclusion Criteria:

* Uterine scar other than low segment cesarean section ( s/p myomectomy, S/p T scar)
* Morbidly adherent placenta during pregnancy
* Cesarean hysterectomy
* Uterine anomaly

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 282 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of uterine niche | Estimated time of two years
  Based on uterine scar measurement -indentation at the site of the cesarean scar with a depth of at least 2 mm

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr Sasson, M.D, Principal Investigator — Sheba Medical Center, Tel-Hashomer
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van der Voet LF, Bij de Vaate AM, Veersema S, Brolmann HA, Huirne JA. Long-term complications of caesarean section. The niche in the scar: a prospective cohort study on niche prevalence and its relation to abnormal uterine bleeding. BJOG. 2014 Jan;121(2):236-44. doi: 10.1111/1471-0528.12542. PMID 24373597
- [Result] Naji O, Abdallah Y, Bij De Vaate AJ, Smith A, Pexsters A, Stalder C, McIndoe A, Ghaem-Maghami S, Lees C, Brolmann HA, Huirne JA, Timmerman D, Bourne T. Standardized approach for imaging and measuring Cesarean section scars using ultrasonography. Ultrasound Obstet Gynecol. 2012 Mar;39(3):252-9. doi: 10.1002/uog.10077. PMID 21858885
- [Result] Roberge S, Boutin A, Chaillet N, Moore L, Jastrow N, Demers S, Bujold E. Systematic review of cesarean scar assessment in the nonpregnant state: imaging techniques and uterine scar defect. Am J Perinatol. 2012 Jun;29(6):465-71. doi: 10.1055/s-0032-1304829. Epub 2012 Mar 7. PMID 22399223
- [Result] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016
- [Result] Wang CB, Chiu WW, Lee CY, Sun YL, Lin YH, Tseng CJ. Cesarean scar defect: correlation between Cesarean section number, defect size, clinical symptoms and uterine position. Ultrasound Obstet Gynecol. 2009 Jul;34(1):85-9. doi: 10.1002/uog.6405. PMID 19565535
- [Result] Osser OV, Jokubkiene L, Valentin L. Cesarean section scar defects: agreement between transvaginal sonographic findings with and without saline contrast enhancement. Ultrasound Obstet Gynecol. 2010 Jan;35(1):75-83. doi: 10.1002/uog.7496. PMID 20034000